CLINICAL TRIAL: NCT05268263
Title: Evaluating the Feasibility of Artificial Intelligence Algorithms in Clinical Settings for Classification of Normal, Wheeze and Crackle Sounds Acquired From a Digital Stethoscope
Brief Title: Feasibility of AI-based Classification of Normal, Wheeze and Crackle Sounds From Stethoscope in Clinical Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innova Smart Technologies (Pvt.) Ltd (Other)
Collaborators: Lady Reading Hospital, Pakistan (Other Government); NOABIO LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pulmo AI LRH
Record Dates: First submitted 2022-01-08; First posted 2022-03-07 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Respiratory; Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Artificial Intelligence Algorithm — The enrolled population will include patients with a history of lung pathologies. Artificial intelligence-based models are developed for classification of wheezes, crackles and normal lung sounds. These AI models will be tested and assessed on local lung sounds clinical data.

SUMMARY:
Assessing the feasibility and testing the accuracy of the developed artificial intelligence algorithms for detection of wheezes and crackles in patients with lung pathologies in clinical settings on unseen local patient data acquired through three digital stethoscopes.

ELIGIBILITY:
Inclusion Criteria:

* Ages all
* Written consent provided

Exclusion Criteria:

* Subject condition unstable
* Chest wall deformity or wounds in adhesive application areas
* Written consent not provided

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Testing the accuracy of artificial intelligence models for detection of wheeze, crackles, and normal lung sounds by measuring the sensitivity and specificity | 2 months
  Artificial intelligence models are trained on lung sounds collected from three different digital stethoscopes named NoaScope, eSteth, and Littmann individually. Data from all three digital stethoscopes is also merged to train separate AI models. These trained AI models will be evaluated based on sensitivity which is the ability to correctly identify wheezes and crackles, and specificity which is the ability to correctly identify normal lung sounds. True positive (TP), true negative (TN), false positive (FP), and false-negative (FN) values will be used to calculate sensitivity & specificity using the following expressions.
  Sensitivity: TP/TP+FN Specificity: TN/TN+FP
Clinical validation of AI models for detection of wheeze, crackles, and normal lung sounds by comparison with gold standard | 2 months
  AI models will be tested for their clinical feasibility through comparison of results obtained from AI models with that of the gold standard by measuring positive and negative agreement (NPA & PPA). The gold standard is the label given to each lung sound recording by an experienced consultant pulmonologist. The AI model is blinded to these labels and is tested independently for detection of normal lung sounds, wheezes, and crackles

SECONDARY OUTCOMES:
Performance analysis of three digital stethoscopes: Littmann, NoaScope, and eSteth | 2 months
  Performance analysis of three digital stethoscopes NoaScope, eSteth, and Littmann will be evaluated using the sensitivity and specificity achieved by each stethoscope. True positive (TP), true negative (TN), false positive (FP), and false-negative (FN) values will be used to calculate sensitivity & specificity using the following expressions.
  Sensitivity: TP/TP+FN Specificity: TN/TN+FP

CONTACTS AND LOCATIONS:
Locations (1):
- Lady Reading Hospital, Pakistan, Peshawar, Pakistan

IPD SHARING:
Plan to Share IPD: No